CLINICAL TRIAL: NCT06297148
Title: Self-management Program for Greater Trochanteric Pain Syndrome: a Randomized Controlled Trial
Brief Title: The HIP Self-management Study
Acronym: HIPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Oslo Metropolitan University (Other); Fysiofondet (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Marianne Bakke Johnsen, Principal investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/590816
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: GTPS - Greater Trochanteric Pain Syndrome; Gluteal Tendinopathy; Trochanteric Bursitis; Lateral Hip Pain
Keywords: Greater Trochanteric Pain Syndrome; Lateral hip pain; Gluteal tendinopathy; Trochanteric bursitis; Self-management
MeSH Terms: interventions — Self-Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-management (Experimental): The intervention will consist of 3-5 individual sessions over 12 weeks with a physiotherapist.
  There will be 3 physiotherapists delivering the self-management intervention.
  Interventions: Other: Self-management
- Usual care (Active Comparator): Given standardized information at baseline and free to choose further treatment in primary care.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Self-management — Patients will have 3-5 sessions with a physiotherapist that include individually tailored education, and address physical, cognitive, and behavioral factors deemed as relevant according to the participant's concerns and challenges. Important aspects in this are: problem-solving, decision-making, resource utilization, therapeutic alliance and taking action (The 5 core skills of self-management). SMART goals and an activity plan between sessions will be used as an exposure to maintain, change, or create health behavior.
  Participants will have access to study material, including exercise alternatives and a podcast.
  Arms: Self-management
Other: Usual care — Usual care at the department consists of general information about the condition and advice on pain management and exercise. For further treatment, patients are referred to primary care. Participation in the study will not affect how this is conducted.
  Arms: Usual care

SUMMARY:
The HIPS-study will be an observer blinded, single-centre, parallel-group randomized controlled trial (RCT).

The main purpose of the study is:

1. To investigate the clinical effectiveness of a self- management program versus usual care for patients with greater trochanteric pain syndrome (GTPS).

   * H0: There is no difference between a self-management program and usual care on pain and function in patients with GTPS.
   * H1: There is a difference between a self-management program and usual care on pain and function in patients with GTPS.
2. To investigate if self-management is more cost-effective than usual care in the treatment of patients with GTPS.

Participants will be randomly allocated into one of two groups: 1) self-management program or 2) usual care.

Follow-up will be at 3-, 6- and 12-months.

DETAILED DESCRIPTION:
Background:

Continuous or intermittent lateral hip pain, also known as greater trochanteric pain syndrome (GTPS), is a common chronic and disabling musculoskeletal condition. It usually occurs during the fourth to sixth decades of life, predominantly among women. The prevalence and incidence rates have been reported to be 4.2 and 3.3 per 1000 person-years, respectively, in the general practice population. The impact of GTPS is reported to be debilitation, as it typically disturbs sleep and limits daily function and participation in work.

Exercise and education are considered the cornerstone of treatment, and in recent randomized controlled trials this combination has demonstrated significant improvements in pain and function. However, studies have failed to show any difference between specific hip exercises and non-specific (sham) exercises in combination with patient education. As GTPS is recurrent and persistent of nature, person-centered care and the incorporation of self-management strategies could be beneficial. To the investigators knowledge, this study will be the first one to investigate self-management for the current patient population. Results from the study may change the type, delivery, and content of treatment for patients with GTPS, relevant for both primary- and secondary care.

The main objective of the study is to evaluate the clinical effectiveness of a self-management program compared to usual care for patients with GTPS.

Methods and analyses:

110 patients will be recruited and randomly allocated into one of two groups: 1) self-management or 2) usual care. The randomization sequence will be computer-generated with blocks of various size, unknown to any of the research team. Due to the nature of therapeutic studies, blinding of the participants and the treating physiotherapist is not possible. The investigator assessing the outcome measures will be blinded to group allocation.

Descriptive statistics will be collected at baseline, and presented as means with standard deviation (SD) or as medians with inter quartile range (IQR). The primary analysis will be conducted on the intention to treat population and compare the two intervention groups (self-management vs usual care) on mean difference in pain and disability (VISA-G-N score) at baseline, 3 and 6 months. The estimated mean difference between groups at 6 months (main endpoint) will be analyzed using a longitudinal mixed effects model analysis of covariance. Baseline score on VISA-G-N, time, intervention and interaction between time and intervention will be included as covariates. Secondary outcomes assessed at multiple time points (baseline, 3, 6 and 12 months) will be analyzed by the same approach as described for the primary outcome, on both the intention to treat population and the per protocol population.

The degree of missingness will be explored using sensitivity analysis with multiple imputation and/or the use of an alternative repeated measures mixed model analysis accordingly, to assess the robustness of data. In addition, multivariable logistic and linear regression analysis will be used to explore predictive factors, such as demographics, expectations, clinical findings, and psychosocial factors for primary and secondary outcomes. Model building will be done in a way that is appropriate for the given sample sizes, by restricting the number of potential predictive factors and considering shrinkage methods to stabilize predictions. Mediation analysis will be performed to explore the causal pathway between treatment allocation and the primary outcome of pain and disability by considering, amongst others, pain self-efficacy and emotional distress as potential mediators that may be part of the causal pathway between intervention and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18 and 70 years of age
* History of lateral hip pain > 3 months
* Reported average pain intensity the last week ≥ 3 on a numeric rating scale
* Lateral hip pain is the main complaint
* Pain on palpation of the greater trochanter region
* In addition, lateral hip pain on at least one of the following tests:

  * Single leg stance test: standing 30 seconds on the affected leg
  * FADER: passive stretch/compression of gluteus medius/minimus
  * FADER-R: static muscle test with resistance to internal hip rotation
  * ADD: passive stretch to hip adduction in sidelying
  * ADD-R: resisted hip abduction in sidelying
  * FABER (Patrick's) test

A positive test is defined as a spontaneous reproduction of the participant's lateral hip pain. In participants with bilateral lateral hip pain, the worst hip will be included, and the presence of bilateral pain will be documented.

Exclusion Criteria:

* Significant back pain causing referred pain to the lateral hip
* Clinical signs of radiculopathy
* Symptomatic osteoarthritis
* Other hip joint pathologies
* History of trauma or surgery on the affected side
* Pregnancy or post-partum pelvic pain (under 12 months since birth)
* Active cancer
* Not able to write, read, and comprehend Norwegian (without the use of an interpreter)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute of Sport Assessment Gluteal Questionnaire (VISA-G) | Baseline, 3 months, 6 months, 12 months
  Pain and function. Total score ranges from 0-100, with higher scores representing less pain and disability.

SECONDARY OUTCOMES:
Numeric rating scale (NRS) | Baseline, 3 months, 6 months, 12 months
  Pain intensity (at rest and during activity) during the last week rated on a scale ranging from 0 (no pain) to 10 (worst possible pain).
Painful sites | Baseline, 3 months, 6 months, 12 months
  The number of painful sites (during the last 14 days) divided into 18 anatomical regions. Number of painful sites are added up to give a total score.
The Pain Self-Efficacy Questionnaire (PSEQ) | Baseline, 3 months, 6 months, 12 months
  Confidence in performing activities while in pain. Includes 10-items, where patients rate their confidence from 0 points (not at all confident) to 6 points (completely confident). Total scores are calculated by summing the individual items with a range from 0 points (less self-efficacy) to 60 points (more self-efficacy).
EuroQoL-5 dimensions-5 Level (Eq-5D-5L) | Baseline, 3 months, 6 months, 12 months
  Generic health related quality of life. The first part is based on 5 questions which are answered on a 5-step scale. It gives an index between 0-1, with a higher index representing better quality of life. The second part, EQ-VAS is a vertical line in which the participants mark the point best describing their quality of life. The score ranges from 0-100, where 100 represents best and 0 worst imaginable health states.
Hopkins Symptoms checklist-10 (HSCL-10) | Baseline, 3 months, 6 months, 12 months
  Psychological distress measured on a scale from 1 (not at all) to 4 (extremely). The mean score is calculated producing a range of scores from 1-4 where higher score corresponds to more psychological distress.
iMTA Medical Consumption Questionnaire (iMCQ) | Baseline, 3 months, 6 months, 12 months
  Medical consumption and healthcare utilization. Not measured on a scale, but as total costs. This is estimated based on unit costs collected from national pricelists.
iMTA Productivity Cost Questionnaire (iPCQ) | Baseline, 3 months, 6 months, 12 months
  The costs of productivity loss (absenteeism) are valued in hours, and can be translated by a standard cost price of productivity per hour.
Expectations related to VISA-G | Baseline
  Expected change in pain and function (from baseline to 6 months) related to VISA-G. Total score ranges from 0-100, with higher scores representing less pain and disability.
Expectations on numeric rating scale (NRS) | Baseline, 3 months, 6 months
  Expected change in function and pain rated on a scale from 0 (no pain/full function) to10 (worst possible pain/function)
Global rating of change (GROC) | 6 months
  Perceived change in lateral hip pain from baseline to follow-up at 6 months, measured on an 11-point likert scale ranging from -5 (much worse) to 5 (completely recovered)
Patient acceptable symptom state (PASS) | 6 months
  Patient satisfaction with current symptom state, by asking the question: "Taking into account all the activities you have during your daily life, your level of hip pain, and also your functional impairment, do you consider that your current state is satisfactory?" The response options are "yes" or "no"

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Ullevål, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, that underlie the results reported in the study, will be available to interested researchers upon reasonable request. Proposals should be directed to the data custodian, principal investigator at mamari@oslomet.no.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following publication.
Access Criteria: To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Morin Melas T, Bjorneboe J, Juel NG, Wefring ML, Skatteboe S, Killingmo RM, Engebretsen KB, Rathleff MS, Oiestad BE, Soberg HL, Pripp AH, Brox JI, Johnsen MB. Self-management versus usual care for greater trochanteric pain syndrome (the HIPS trial): study protocol for a randomised controlled trial. BMJ Open. 2025 Apr 5;15(4):e090688. doi: 10.1136/bmjopen-2024-090688. PMID 40187788
- See also: Grimaldi A, Mellor R, Hodges P, Bennell K, Wajswelner H, Vicenzino B. Gluteal Tendinopathy: A Review of Mechanisms, Assessment and Management. Sports Med 2015;45(8):1107-19. (In eng). DOI: 10.1007/s40279-015-0336-5 — https://pubmed.ncbi.nlm.nih.gov/25969366/
- See also: Pianka MA, Serino J, DeFroda SF, Bodendorfer BM. Greater trochanteric pain syndrome: Evaluation and management of a wide spectrum of pathology. SAGE Open Med 2021;9:20503121211022582. (In eng). DOI: 10.1177/20503121211022582 — https://pubmed.ncbi.nlm.nih.gov/34158938/
- See also: Klontzas ME, Karantanas AH. Greater trochanter pain syndrome: a descriptive MR imaging study. Eur J Radiol 2014;83(10):1850-5. (In eng). DOI: 10.1016/j.ejrad.2014.06.009. — https://pubmed.ncbi.nlm.nih.gov/25043986/
- See also: Fearon AM, Scarvell JM, Neeman T, Cook JL, Cormick W, Smith PN. Greater trochanteric pain syndrome: defining the clinical syndrome. Br J Sports Med 2013;47(10):649-53. (In eng). DOI: 10.1136/bjsports-2012-091565. — https://pubmed.ncbi.nlm.nih.gov/22983121/
- See also: Lievense A, Bierma-Zeinstra S, Schouten B, Bohnen A, Verhaar J, Koes B. Prognosis of trochanteric pain in primary care. Br J Gen Pract 2005;55(512):199-204. (In eng). — https://pubmed.ncbi.nlm.nih.gov/15808035/
- See also: Plinsinga ML, Coombes BK, Mellor R, et al. Psychological factors not strength deficits are associated with severity of gluteal tendinopathy: A cross-sectional study. Eur J Pain 2018;22(6):1124-1133. (In eng). DOI: 10.1002/ejp.1199. — https://pubmed.ncbi.nlm.nih.gov/29427310/
- See also: Stephens G, O'Neill S, Mottershead C, Hawthorn C, Yeowell G, Littlewood C. "It's just like a needle going into my hip, basically all of the time". The experiences and perceptions of patients with Greater Trochanteric Pain syndrome in the UK National Hea — https://pubmed.ncbi.nlm.nih.gov/32452392/
- See also: Stephens G, O'Neill S, French HP, et al. A survey of physiotherapy practice (2018) in the United Kingdom for patients with greater trochanteric pain syndrome. Musculoskelet Sci Pract 2019;40:10-20. (In eng). DOI: 10.1016/j.msksp.2019.01.004. — https://pubmed.ncbi.nlm.nih.gov/30660989/
- See also: French HP, Woodley SJ, Fearon A, O'Connor L, Grimaldi A. Physiotherapy management of greater trochanteric pain syndrome (GTPS): an international survey of current physiotherapy practice. Physiotherapy 2020;109:111-120. (In eng). DOI: 10.1016/j.physio.20 — https://pubmed.ncbi.nlm.nih.gov/31493863/
- See also: Cowan RM, Ganderton CL, Cook J, Semciw AI, Long DM, Pizzari T. Does Menopausal Hormone Therapy, Exercise, or Both Improve Pain and Function in Postmenopausal Women With Greater Trochanteric Pain Syndrome? A 2 × 2 Factorial Randomized Clinical Trial. Am — https://pubmed.ncbi.nlm.nih.gov/34898293/
- See also: Ganderton C, Semciw A, Cook J, Moreira E, Pizzari T. Gluteal Loading Versus Sham Exercises to Improve Pain and Dysfunction in Postmenopausal Women with Greater Trochanteric Pain Syndrome: A Randomized Controlled Trial. J Womens Health (Larchmt) 2018;27( — https://pubmed.ncbi.nlm.nih.gov/29715073/
- See also: Mellor R, Bennell K, Grimaldi A, et al. Education plus exercise versus corticosteroid injection use versus a wait and see approach on global outcome and pain from gluteal tendinopathy: prospective, single blinded, randomised clinical trial. Br J Sports — https://pubmed.ncbi.nlm.nih.gov/30385462/
- See also: Kjeldsen T, Hvidt KJ, Bohn MB, et al. Exercise compared to a control condition or other conservative treatment options in patients with Greater Trochanteric Pain Syndrome: a systematic review and meta-analysis of randomized controlled trials. Physiother — https://pubmed.ncbi.nlm.nih.gov/38295551/
- See also: Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med 2003;26(1):1-7. (In eng). DOI: 10.1207/s15324796abm2601_01. — https://pubmed.ncbi.nlm.nih.gov/12867348/

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT06297148/SAP_002.pdf